CLINICAL TRIAL: NCT06135259
Title: Topical Erythropoietin Hydrogel in Management of Oral Lichen Planus: A Randomized Controlled Clinical Trial
Brief Title: Topical Erythropoietin Hydrogel in Management of Oral Lichen Planus
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FDASU-RecIR022222
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2023-04

CONDITIONS: Oral Lichen Planus
Keywords: erythropoietin gel; tumor necrosis factor; oral lichen planus
MeSH Terms: conditions — Lichen Planus, Oral | interventions — Erythropoietin; Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- erythropoietin mucoadhesive thermosensitive hydrogel (Experimental): erythropoietin solutions of 150, 300, and 500 IU/mL were mixed with trimethyl chitosan (M) solutions. glycerophosphate solution was then added to the mixture to obtain erythropoietin-loaded hydrogel comprising final concentrations of trimethyl chitosan (5%) and glycerophosphate (20%).
  Interventions: Drug: erythropoietin
- Triamcinolone Mucoadhesive gel (Active Comparator): Each 0.1 mg triamcinolone acetonide in a dental paste containing gelatin, pectin, cream flavor, vanilla flavor and carboxymethylcellulose sodium in Plasticized Hydrocarbon Gel, a polyethylene and mineral oil gel base.
  Interventions: Drug: Triamcinolone acetonide

INTERVENTIONS:
Drug: erythropoietin — erythropoietin solutions of 150, 300, and 500 IU/mL were mixed with trimethyl chitosan (M) solutions. glycerophosphate solution was then added to the mixture to obtain erythropoietin-loaded hydrogel comprising final concentrations of trimethyl chitosan(5%) and glycerophosphate (20%).
  Other Names: erythropoietin mucoadhesive thermosensitive hydrogel
  Arms: erythropoietin mucoadhesive thermosensitive hydrogel
Drug: Triamcinolone acetonide — Each 0.1 mg triamcinolone acetonide in a dental paste containing gelatin, pectin, cream flavor, vanilla flavor and carboxymethylcellulose sodium in Plasticized Hydrocarbon Gel, a polyethylene and mineral oil gel base.
  Other Names: Triamcinolone Mucoadhesive gel
  Arms: Triamcinolone Mucoadhesive gel

SUMMARY:
The purpose of this study is to compare the clinical efficacy of erythropoietin gel containing a solution of 4000 units with triamcinolone acetonide 0.1% gel in the treatment of symptomatic oral lichen planus (OLP)

DETAILED DESCRIPTION:
At the first visit before the initiation of the study;

* Information including age, gender, disease process, medical history, drug history, family history, and clinical symptoms and signs will be documented.
* Patients will be examined clinically by magnifying mirror using a spotlight for the oral lesions, the distribution of the lesions and the affected areas will be recorded, and a punch biopsy will be taken to confirm the diagnosis.

Twenty-four patients seeking treatment for symptomatic OLP will be assessed for eligibility for this study. Patients will be recruited from the outpatient clinic, department of Oral Medicine and Periodontology, Faculty of Dentistry, and the Department of Skin and Venereal Disease, Faculty of Medicine, Ain Shams University.

The study will be conducted according to the ethical principles provided by the Declaration of Helsinki and according to the principles of good clinical practice. Faculty of Dentistry-Ain Shams University Research Ethical Committee (FD-ASU-RECD) will review the protocol, the procedure will be fully explained to the patients. Each patient will receive detailed verbal and written information about the study protocol. Understanding and agreement to enroll in the study will be confirmed and written consent forms will be obtained.

II- Study design, interventions, blinding, randomization, and grouping:

The study is designed as a Randomized- parallel 2 arm - assessor blinded single center- controlled comparative clinical trial with immunohistochemical analysis.

* Interventions The oral Gel carrier of the intervention will be designed, prepared, and in vitro characterized at the Pharmaceutical Science Department, Faculty of Pharmacy- Ain University.
* Patients grouping Patients who met the eligibility criteria will be randomly assigned to 2 different treatment regimens using computer-generated random tables and allocation concealment;

Group I Will include twelve patients with oral lichen planus lesions receiving ( erythropoietin mucoadhesive thermosensitive hydrogel), twice daily (Experimental Arm)

Group II:

It will include twelve patients with oral lichen planus lesions receiving (Topical corticosteroid 0.1%) four times per day for 8 weeks (Positive control arm) In the fourth- and eighth both patients in group II will receive topical antifungal (Miconazole 2%) to avoid secondary candidiasis while patients in group I will receive topical antifungal only if needed

ELIGIBILITY:
Inclusion Criteria:

1. Clinically proven painful symptomatic forms of OLP confirmed by the presence of red or erythematous changes, or shallow ulcerations with fine lacy lines at the periphery of the lesion accentuated by stretching and not eliminated by rubbing (Wickham's striae)
2. Histopathological proven symptomatic OLP

Exclusion Criteria:

1. History of the drug-induced lichenoid lesion.
2. Presence of systemic conditions as; serious active or recurrent infections, malignancy, diabetes mellitus, hypertension, or significant heart, liver, or renal diseases. Assessed using a medical questionnaire guided by the Cornell Medical Index
3. Smoking
4. Known hypersensitivity or severe adverse effects to the treatment drugs or to any ingredient of their preparation as mentioned in history
5. Pregnancy or breastfeeding.
6. History of previous treatments potentially effective on OLP such as antimalarial agents, retinoids, corticosteroids, or immunosuppressive drugs from less than 2 weeks for topical medications, and 4 weeks for systemic medications before starting the study
7. Loss of pliability or flexibility in the tissues involved by the lesions of OLP.
8. Histological signs of epithelial dysplasia or lichenoid lesions within the biopsied sites.
9. Patients with extensive skin lesions and indicated for systemic corticosteroids.
10. Vulnerable groups (Handicapped, orphans, or prisoners)

    -

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-05-20 (Estimated); Primary Completion 2024-07-23 (Estimated); Study Completion 2024-09-23 (Estimated)

PRIMARY OUTCOMES:
Clinical Scoring | The assessment will be carried out at baseline, 1 month and 2 months after starting the treatment protocol and then at 3 months after the end of the observational period
  The marker lesion in each patient will be assessed for areas of reticulation, erosion, and ulceration by visual examination and the scoring will be recorded as follow:
  0: Mild represented no lesion/normal mucosa.
  1. White striae/no erythematous area.
  2. White striae with atrophic area less than 1 cm2
  3. White striae with atrophic area of more than 1 cm2
  4. White striae with an erosive area less than 1 cm2
  5. White striae with an erosive area of more than 1cm2
Visual Analogue Score | The assessment will be carried out at baseline, 1 month and 2 months after starting the treatment protocol and then at 3 months after the end of the observational period
  The Visual Analogue Score consisted of a 10-cm horizontal line marked 0-10 (0 no pain; 10 most severe pain experienced). Patients will mark the scale at each visit. The Visual Analogue Score is then scored by measuring from the patient's mark to the beginning of the scale in cm, and all Visual Analogue Score will be included on one sheet of paper allowing the patient to think in terms of change instead of absolutes.
Imaging and measuring surface area of the oral lesion | The assessment will be carried out at baseline, 1 and 2 months after starting the treatment protocol and then at 3 months after the end of the observational period
  Standardized photographs of the oral marker lesion for each patient will be taken with the same digital camera and setting, and the surface area of the lesion will be outlined and measured using specific image software.

SECONDARY OUTCOMES:
Tumor necrosis factor Salivary level | The Salivary Sample for each patient will be taken at baseline and after 2 months treatment period.
  The patient will export 10 ml of unstimulated whole saliva into a sterile centrifuge.
  tube. The saliva will be centrifuged, filtered, and frozen until use. The mean concentration of TNF-α in the whole saliva of in patients with OLP lesions will be measured by ELISA kit. The assay will be performed according to the manufacturer's instruction The patient will export 10 ml of unstimulated whole saliva into a sterile centrifuge.
  tube. The saliva will be centrifuged, filtered, and frozen until use. The mean concentration of TNF-α in the whole saliva of in patients with OLP lesions will be measured by ELISA kit. The assay will be performed according to the manufacturer's instruction

CONTACTS AND LOCATIONS:
Overall Officials: Yasmine A Fouad, Ph.D, Principal Investigator — Ain Shams University